CLINICAL TRIAL: NCT00978861
Title: A Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate of The Whitening Efficacy and Safety of REMEWHITE
Brief Title: Clinical Study to Evaluate of The Whitening Efficacy and Safety of REMEWHITE
Acronym: REMEWHITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JDC Tech (Industry)
Responsible Party: Je-Uk park / PI, The catholic university of korea seoul st. mary's hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RE5
Record Dates: First submitted 2009-08-31; First posted 2009-09-17 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Tooth Whitening
MeSH Terms: interventions — Hydrogen Peroxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- whitening (Experimental): 30% Hydrogen peroxide
  Interventions: Drug: Hydrogen Peroxide

INTERVENTIONS:
Drug: Hydrogen Peroxide — Whitening product syringe type

SUMMARY:
The purpose of this study is to determine the effect of REMEWHITE on tooth whitening.

DETAILED DESCRIPTION:
This study intended to establish the efficacy of REMEWHITE after using the product under controlled conditions at the hospital.

The efficacy of the product was assessed at the end of the study; clinical examination by the dentist.

ELIGIBILITY:
Inclusion Criteria:

* ability to understand and provide informed consent
* general good health male and female adults, were 20 years or older
* no pregnant woman
* had six caines-free maxillary anterior teeth without restorations on the labial surfaces

Exclusion Criteria:

* had severe internal discoloration (tetracycline stains, fluorosis, pulpless teeth)
* evidence of fracture or major cracks on tooth
* were pregnant or nursing
* had tooth sensitivity
* smokers
* had teeth shade A1, A2

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
colorimeter | 12 weeks after treatment

SECONDARY OUTCOMES:
colorimeter | 24 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Je-Uk Park, PI, Principal Investigator — The cathiloc university of korea seoul st. mary's hospital
Locations (1):
- The cathiloc university of korea seoul st. mary's hospital, Seoul, South Korea